CLINICAL TRIAL: NCT00937651
Title: Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Antihypertensive Efficacy, Safety, Tolerability, and Pharmacodynamic/Pharmacokinetic Profiles After 4 Weeks of Oral Administration of Fimasartan(BR-A-657) at 20-180mg in Patients With Essential Hypertension
Brief Title: Efficacy, Safety and Pharmacodynamic/Pharmacokinetic Study of Fimasartan (BR-A-657•K)
Acronym: Fimasartan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Jeongeun / Director, Boryung Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A657-BR-CT-201
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo, 3 tablets
  Interventions: Drug: Placebo
- BR-A-657•K 20 mg group (Active Comparator): Fimasartan 20 mg, 1 tablet + placebo, 2 tablets
  Interventions: Drug: Fimasartan (BR-A-657•K) 20 mg
- BR-A-657•K 60 mg group (Active Comparator): Fimasartan 20 mg, 1 tablet + 40 mg, 1 tablet + placebo 1 tablet
  Interventions: Drug: Fimasartan (BR-A-657•K) 60 mg
- BR-A-657•K 180 mg group (Active Comparator): Fimasartan 20 mg, 1 tablet + 80 mg, 1 tablet + 80 mg 1 tablet
  Interventions: Drug: Fimasartan (BR-A-657•K) 180 mg

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Fimasartan (BR-A-657•K) 20 mg — Fimasartan 20 mg, 1 tablet + placebo, 2 tablets
  Other Names: Fimasartan
  Arms: BR-A-657•K 20 mg group
Drug: Fimasartan (BR-A-657•K) 60 mg — Fimasartan 20 mg, 1 tablet + 40 mg, 1 tablet + placebo 1 tablet
  Other Names: Fimasartan
  Arms: BR-A-657•K 60 mg group
Drug: Fimasartan (BR-A-657•K) 180 mg — Fimasartan 20 mg, 1 tablet + 80 mg, 1 tablet + 80 mg 1 tablet
  Other Names: Fimasartan
  Arms: BR-A-657•K 180 mg group

SUMMARY:
Study objective:

1. To evaluate the antihypertensive efficacy, safety and tolerability of the drug after the oral administration of BR-A-657•K at 20~180mg for 4 weeks to patients with essential hypertension.
2. To review the pharmacokinetic profile after the multiple administration and the pharmacodynamic profile regarding the renin-angiotensin system, after the oral administration of BR-A-657•K at 20~180mg for 4 weeks to patients with essential hypertension.
3. To determine the dose for the clinical study at the next phase by analyzing the relationship between the antihypertensive efficacy and pharmacokinetic • pharmacodynamic results.

DETAILED DESCRIPTION:
Fimasartan (BR-A-657-K), a selective blocker of AT1 receptor subtype, showed the rapid and potent antihypertensive effect in many hypertensive models. Phase I study, Fimasartan (BR-A-657-K) 20mg ~ 480mg single dosing with healthy subjects, demonstrated that the Fimasartan (BR-A-657-K) was very safe and well tolerated. Another phase I study, Fimasartan (BR-A-657-K) 120mg and 360mg dosing for 7 days, also showed that Fimasartan (BR-A-657-K) was safe and tolerable though one temporal adverse event was observed in high dose.

A randomized, double-blind, placebo-controlled, parallel grouped, clinical study will be conducted to evaluate the antihypertensive efficacy and tolerability and to determine adequate antihypertensive dosage of Fimasartan(BR-A-657-K) in patients with mild to moderate essential hypertension.

Approximately 60 patients will be enrolled over 12 months in Seoul National University Hospital.

After 2 weeks of placebo run-in period, all subjects will be randomized into one of the following 5 groups. Subjects will take test drug/placebo for 28 days of treatment period. If subjects take any antihypertensive medications before screening, the subjects will have 1 week of wash-out period.

Group I : Placebo, Group II : Fimasartan 20 mg, Group III: Fimasartan 60 mg, Group IV : Fimasartan 180 mg

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women, aged 18 - 65
* Patients with mild to moderate essential hypertension: On both screening and Day -1 visit, mean sitting DBP should be ≥ 95mmHg and ≤ 114mmHg, and ΔDBP on Day -14 and Day -1 should be within 7 mmHg
* Patients who gave their consent to participate in this study and signed the written informed consent form
* Patients who have understood the study, and been judged to be cooperative and able to participate in the study until the study completion date

Exclusion Criteria:

1. Women of childbearing potential who have not received the hysterectomy or men who are not willing to use birth control measures.
2. Patients whose sitting DBP is < 95mmHg or ≥ 115mmHg. Patients with severe hypertension whose SBP is ≥200mmHg
3. Patients with secondary hypertension
4. Patients with severe renal disease, gastrointestinal disorder, hematologic disorder, liver disease, etc. that can affect the absorption, distribution, metabolism and excretion of drugs
5. Patients with symptoms of orthostatic hypotension
6. Patients with severe insulin dependent diabetes or uncontrolled diabetes
7. Patients who suffered myocardial infarction or serious coronary arterial disease over the past 6 months or patients with clinically significant congestive heart failure or valvular heart disease
8. Patients with consumption disease, autoimmune disease, or connective tissue disease
9. Patients with the history of type B hepatitis or type C hepatitis
10. Patients with HIV infection or hepatitis
11. Patients with clinically significant abnormal laboratory test findings
12. Patients on any drug treatment that might affect the blood pressure
13. Patients with allergy or contraindication to angiotensin II-receptor antagonists
14. Patients with current or suspected alcohol addiction or history of drug abuse
15. Patients whose mean weight lies out of the range of -15% ~ +35%, based on the Modified Metropolitan Life Insurance table
16. Patients who are not eligible as subjects of the study, as determined by the principal investigator or a sub-investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
the level of sitting diastolic blood pressure reduction | Day -1 vs Day 27

SECONDARY OUTCOMES:
the level of sitting systolic blood pressure reduction, mean blood pressure (MBP), 24-hr day-time, night-time SBP and DBP, T/P ratio based on the 24-hr Ambulatory Blood Pressure Monitoring | Day -1 vs Day 27

REFERENCES:
- [Derived] Lee H, Yang HM, Lee HY, Kim JJ, Choi DJ, Seung KB, Jeon ES, Ha JW, Rim SJ, Park JB, Shin JH, Oh BH. Efficacy and tolerability of once-daily oral fimasartan 20 to 240 mg/d in Korean Patients with hypertension: findings from Two Phase II, randomized, double-blind, placebo-controlled studies. Clin Ther. 2012 Jun;34(6):1273-89. doi: 10.1016/j.clinthera.2012.04.021. Epub 2012 May 17. PMID 22608107